CLINICAL TRIAL: NCT03116516
Title: A Randomized, Open-label, Single Dose, Crossover Clinical Trial to Compare the Safety and Pharmacokinetics of YHP1604 in Comparison to the Co-administration of Telmisartan/Amlodipine and Rosuvastatin in Healthy Volunteers
Brief Title: Clinical Trial to Compare the Safety and Pharmacokinetics of YHP1604 in Comparison to the Co-administration of Telmisartan/Amlodipine and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP1604-102
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, single dose, crossover clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM1 (Other): In ARM1, 30 subjects will be assigned and the subjects will be administered "telmisartan/amlodipine and rosuvastatin" at Day1 and "YHP1604" at Day22.
  Interventions: Drug: Temisartan/Amlodipine+Rosuvastatin; Drug: YHP1604
- ARM2 (Other): In ARM2, 30 subjects will be assigned and the subjects will be administered "YHP1604" at Day1 and "telmisartan/amlodipine and rosuvastatin" at Day22.
  Interventions: Drug: Temisartan/Amlodipine+Rosuvastatin; Drug: YHP1604

INTERVENTIONS:
Drug: Temisartan/Amlodipine+Rosuvastatin — All subjects will receive a single oral dose of temisartan/amlodipine+rosuvastatin administered in the morning.
  Other Names: Twynsta Tab.+Crestor Tab.
Drug: YHP1604 — All subjects will receive a single oral dose of YHP1604 administered in the morning.
  Other Names: FDC

SUMMARY:
This is a phase 1, open label, single-dose, crossover study to investigate the pharmacokinetics of YHP1604 in comparison to the co-administration of telmisartan/amlodipine and rosuvastatin in healthy male volunteers

Hypothesis: "YHP1604" and "telmisartan/amlodipine and rosuvastatin" are showing equal pharmacokinetics.

DETAILED DESCRIPTION:
This is a phase 1, open label, single-dose, crossover study to investigate the pharmacokinetics of YHP1604 in comparison to the co-administration of telmisartan/amlodipine and rosuvastatin in healthy male volunteers.

In ARM1, 30 subjects will be assigned and the subjects will be administered "telmisartan/amlodipine and rosuvastatin" at Day1 and "YHP1604" at Day22.

In ARM2, 30 subjects will be assigned and the subjects will be administered "YHP1604" at Day1 and "telmisartan/amlodipine and rosuvastatin" at Day22.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male with body mass index(BMI) between 18.5 and 30 kg/m2
* Who has not suffered from clinically significant disease
* Provision of signed written informed consent

Exclusion Criteria:

* History of and clinically significant disease
* A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs
* Administration of other investigational products within 3 months prior to the first dosing
* Volunteers considered not eligible for the clinical trial by the investigator due to reasons including laboratory test results, ECGs, or vital signs

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male with body mass index(BMI) between 18.5 and 30kg/m2
Enrollment: 62 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Telmisartan/Amlodipine/Rosuvastatin Cmax, AUClast | 0 - 72 hrs, 0 - 168 hrs, 0 - 48 hrs
  Cmax, AUClast

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No